CLINICAL TRIAL: NCT06081491
Title: Association Between Molar-Incisor Hypomineralization, Maternal Stress and Anxiety in a Group of Pediatric Patients : A Cross-Sectional Study.
Brief Title: Association Between Molar-Incisor Hypomineralization, Maternal Stress and Anxiety: A Cross-Sectional Study.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sarah Mahmoud Mohamed Sadek, Master student principal investigator, Cairo University
Other Study IDs: MIH and stress
Record Dates: First submitted 2023-10-07; First posted 2023-10-13 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Molar Incisor Hypomineralization
MeSH Terms: conditions — Molar Hypomineralization | interventions — Diagnosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: diagnosis — Pediatric patients within the inclusion criteria will be diagnosed for MIH by the primary investigator and the questionnaire will be filled with face to face interviews with their parents

SUMMARY:
This study aims to evaluate the association between Molar-Incisor Hypomineralization, Maternal Stress and anxiety in a group of pediatric patients.

DETAILED DESCRIPTION:
Molar incisor hypomineralization is a medical global condition characterised by a qualitative defect in the enamel mineralization affecting the first permanent molar teeth predominantly, and with or without the involvement of incisor teeth. MIH have various and major clinical challenges. Clinically the lesion appears with well demarcated opacity and porous with a color that ranges from white, creamy or yellow to brownish. Thus differ in its severity from mild to severe. The OHRQoL is a fundamental part of our children's general health and well-being but with the condition mentioned above their eating, sleeping, social interaction, self-esteem is being minimized and so the analysis of the etiological factors should be carried out.

Worldwide the prevalence of this condition, MIH was found to be from 2.4 to 40%, the reason behind this huge range difference is the use of different indices, diagnostic criteria, variability between examiners, lack of standardized methods of recording lesions and different age groups, while recent studies in Egypt reported 2.3% of MIH in a group of Egyptian children from 8 to 12 years in Cairo. Moreover, 878 million people across the world were MIH-affected and 17.5 million new cases are identified each year according to a study published 02 August 2022 in Egypt.

Despite the worldwide increasing interest in the causes of MIH, there is still insufficient evidence to verify the etiological factors of this condition, especially stress and anxiety. There is a potential relationship between stress and MIH, as glucocorticoids mainly cortisol have receptors on ameloblasts and so further research and population-based studies are urgently required to evaluate the prevalence of MIH and its association with stress.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric Patients with completely erupted at least one first permanent molar with MIH, based on a validated diagnostic criteria
* Children age range from 8 and 12 years
* Parents who agree and signed the consent for their children participation

Exclusion Criteria:

-Enamel defects only limited to the Permanent incisors; as the term MIH was chosen to always highlight the fact that molars are involved regularly in this condition, opacities on incisors only may relate to another origin of the defect and should not be referred to as MIH.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric patients age range of 8 to 12 years with completely erupted at least one first permanent molar and whose parents agree their participation with signed consent will be diagnosed for MIH according to EAPD diagnostic criteria
Sampling Method: Probability Sample
Enrollment: 174 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
MIH occurrence due to stressful events | baseline
  Questionnaire(Brejawi MS etal .2022), Multiple choice questions , (yes or no if yes the participant should choose the degree:not at all/ very little/little/alot) where alot means it has the greatest impact of stress on the child.

CONTACTS AND LOCATIONS:
Overall Officials: Soaad A Moniem, Proffesor, Study Director — Cairo University

REFERENCES:
- [Background] Brejawi MS, Venkiteswaran A, Ergieg SMO, Sabri BM. Correlation between Molar-Incisor Hypomineralization, Stress, and Family Functioning. J Int Soc Prev Community Dent. 2022 Oct 31;12(5):547-553. doi: 10.4103/jispcd.JISPCD_105_22. eCollection 2022 Sep-Oct. PMID 36532319
- See also: Molar Incisor Hypomineralization, Prevalence, and Etiology — https://pubmed.ncbi.nlm.nih.gov/24949012/